CLINICAL TRIAL: NCT02792816
Title: A Multi-site Cohort Observational Study for Molecular Assessment of Artemisinin Resistance Falciparum Malaria in Myanmar
Brief Title: Molecular Surveillance of Artemisinin Resistance Malaria in Myanmar
Status: Completed | Type: Observational
Sponsor: Department of Medical Research, Lower Myanmar (Other)
Collaborators: Kangwon National University (Other)
Responsible Party: Principal Investigator, Myat Htut Nyunt, Research Scientist, Department of Medical Research, Lower Myanmar
Other Study IDs: KMRL_2016_02
Record Dates: First submitted 2016-05-31; First posted 2016-06-08 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Drug Resistance; Plasmodium Falciparum Malaria
MeSH Terms: conditions — Malaria, Falciparum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Finger prick blood samples were taken onto filter paper and Keep dry until DNA extraction.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- Kawthaung Site: The efficacy and safety of the ACT in different sentinel sites will be assessed. The administrated anti-malarial were same and all will be administrated under direct observation. The dosage will be calculated by weight of the patients. Kawthaung is one of the sentinel site and located at the Southern Myanmar.
  Interventions: Drug: First line antimalarial in Myanmar (artemether-lumefrantrine, dihydroartemisinin-piperaquine, and artesunate-mefloquine)
- Myawaddy Site: The efficacy and safety of the ACT in different sentinel sites will be assessed. The administrated anti-malarial were same and all will be administrated under direct observation. The dosage will be calculated by weight of the patients. Myawaddy is one of the sentinel site and located at the northern part of the Southern Myanmar.
  Interventions: Drug: First line antimalarial in Myanmar (artemether-lumefrantrine, dihydroartemisinin-piperaquine, and artesunate-mefloquine)
- Thanbyuzayat Site: The efficacy and safety of the ACT in different sentinel sites will be assessed. The administrated anti-malarial were same and all will be administrated under direct observation. The dosage will be calculated by weight of the patients. Thanbyuzayat is one of the sentinel site and located at the northern part of the Southern Myanmar.
  Interventions: Drug: First line antimalarial in Myanmar (artemether-lumefrantrine, dihydroartemisinin-piperaquine, and artesunate-mefloquine)
- Shwegyin Site: The efficacy and safety of the ACT in different sentinel sites will be assessed. The administrated anti-malarial were same and all will be administrated under direct observation. The dosage will be calculated by weight of the patients. Shwegyin is one of the sentinel site and located at the southern part of the central Myanmar.
  Interventions: Drug: First line antimalarial in Myanmar (artemether-lumefrantrine, dihydroartemisinin-piperaquine, and artesunate-mefloquine)
- Magway Site: The efficacy and safety of the ACT in different sentinel sites will be assessed. The administrated anti-malarial were same and all will be administrated under direct observation. The dosage will be calculated by weight of the patients. Magway is one of the sentinel site and located at the middle part of the central Myanmar.
  Interventions: Drug: First line antimalarial in Myanmar (artemether-lumefrantrine, dihydroartemisinin-piperaquine, and artesunate-mefloquine)
- Rakhine Site: The efficacy and safety of the ACT in different sentinel sites will be assessed. The administrated anti-malarial were same and all will be administrated under direct observation. The dosage will be calculated by weight of the patients. Rakhine is one of the sentinel site and located at the western Myanmar.
  Interventions: Drug: First line antimalarial in Myanmar (artemether-lumefrantrine, dihydroartemisinin-piperaquine, and artesunate-mefloquine)

INTERVENTIONS:
Drug: First line antimalarial in Myanmar (artemether-lumefrantrine, dihydroartemisinin-piperaquine, and artesunate-mefloquine) — Being a observational cohort study, one of the ACT was selected in each study site to assess the efficacy and safety.

SUMMARY:
Efficacy and safety of the artemisinin combination therapy (ACT) in uncomplicated falciparum malaria patients in Myanmar and artemisinin molecular markers analysis

DETAILED DESCRIPTION:
The investigators assessed the efficacy and safety of the ACT in uncomplicated falciparum malaria in different sentinel sites in Myanmar. The recruited patients were follow-up until day 28 or day-42 based on the ACTs. Day-0 samples were analysed for artemisinin molecular markers, (K13 kelch propeller, Pfmdr2, Pffd and Pfarps10).

ELIGIBILITY:
Inclusion Criteria:

* Plasmodium falciparum mono infection by microscopy
* Presence of axillary equal to or more than 37.5 degrees centigrade or history of fever during the past 24 hours
* Ability to swallow oral medication
* Ability and willingness to comply with the study protocol for the duration of the study and to comply with the study visit schedule
* Informed consent from the patient or from a parent or guardian in the case of children

Exclusion Criteria:

* Presence of signs of severe falciparum malaria according to the definitions of World Health Organisation (WHO)
* Mixed or mono-infection with another Plasmodium species detected by microscopy
* Presence of severe malnutrition (defined as a child whose growth standard is below 3 z-score, has symmetrical oedema involving at least the feet or has a mid-upper arm circumference below 110 mm)
* Presence of febrile conditions due to diseases other than malaria (e.g. measles, acute lower respiratory tract infection, severe diarrhoea with dehydration) or other known underlying chronic or severe diseases (e.g. cardiac, renal and hepatic diseases, Human Immune Deficiency Virus (HIV)/Acquired Immune Deficiency Syndrom (AIDS)
* Regular medication, which may interfere with antimalarial pharmacokinetics
* History of hypersensitivity reactions or contraindications to any of the medicine(s) being tested or used as alternative treatment(s)
* A positive pregnancy test or breastfeeding
* Unable to or unwilling to take a pregnancy test or contraceptives

Ages: 3 Months to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study populations were selected purposely based on the previous evidence of the drug resistance in Myanmar
Sampling Method: Non-Probability Sample
Enrollment: 550 (Actual)
Dates: Start 2009-06; Primary Completion 2013-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Proportion of adequate clinical and parasitological response (ACPR) | day 28 or day 42 after initial dose of ACT
  For artesunate-mefloquine or dihydroartemisinin-piperaquine, 42 days follow-ups and for artemether-lumefrantrine combinations, 28 days followe-ups

SECONDARY OUTCOMES:
Proportion of the day-3 parasite positivity after ACT by microscopy | 3rd day after initial dose of ACT
  72 hr after ACT is one of the indicator for delayed clearance of parasitaemia in falciparum malaria
Treatment failure rate | anytime within observation period (28/42 days after treatment with one of ACTs)
  Early Treatment Failure (ETF), Late Clinical Failure (LCF), Late Parasitological Failure (LPF) based on the WHO standard protocol and definitions
Mutant rate | Day-0 samples
  Day-0 samples were used to amplify the artemisinin resistance molecular markers to know the mutant rate in each study sites

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Myat Phone Kyaw, Yangon, Yangon, Burma

IPD SHARING:
Plan to Share IPD: Undecided
We may share the data on request after publication.

REFERENCES:
- [Derived] Nyunt MH, Soe MT, Myint HW, Oo HW, Aye MM, Han SS, Zaw NN, Cho C, Aung PZ, Kyaw KT, Aye TT, San NA, Ortega L, Thimasarn K, Bustos MDG, Galit S, Hoque MR, Ringwald P, Han ET, Kyaw MP. Clinical and molecular surveillance of artemisinin resistant falciparum malaria in Myanmar (2009-2013). Malar J. 2017 Aug 14;16(1):333. doi: 10.1186/s12936-017-1983-9. PMID 28806957